CLINICAL TRIAL: NCT05384054
Title: Association Between Erythroferron and Perioperative Hemoglobin Levels in Patient Undergoing Heart Valve Surgery
Status: Completed | Type: Observational
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Other Study IDs: 4-2022-0260
Record Dates: First submitted 2022-05-09; First posted 2022-05-20 (Actual); Last update posted 2025-10-02 (Actual); Status verified 2025-09

CONDITIONS: Postoperative Anemia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Plasma for Erythroferrone/Hepcidin/FGF-23 measurement
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Lowest Erythroferron tertile group: The lowest concentration group will be Group1.
- Highest Erythroferron tertile group: The highest concentration group will be Group2.

SUMMARY:
In patients undergoing cardiac surgery, perioperative anemia is an important factor in surgical recovery. In addition to the low preoperative hemoglobin level, the delayed recovery of the postoperative hemoglobin level is an important problem affecting the incidence of postoperative anemia. Erythroferron is the early response to of the red blood cell production in stressful situations such as anemia, bleeding, and hypoxia. Therefore, it is thought that acute blood loss and systemic inflammatory reaction that inevitably occurs after cardiac surgery will synthesize erythroferron, which helps to restore hemoglobin level at postoperative period by promoting hematopoiesis by simultaneously inhibiting hepcidin and activating hematopoiesis.

In this study, the investigators will investigate the association between Erythroferron and perioperative hemoglobin levels in patient undergoing heart valve surgery.

ELIGIBILITY:
Inclusion Criteria:

* Patients older than 20 years
* undergoing elective valvular heart surgery

Exclusion Criteria:

* Emergency operation
* Co-operation with other surgeries
* Patients with cardiogenic shock or ventricular-assist device (eg. ECMO, IABP)
* Patients requiring mechanical ventilator care in preoperative period
* Patient with severe chronic kidney disease (GFR(CKD-EPI) <30ml/min/1.73m2)
* Patients with preoperative infection status (Eg. Sepsis)
* Patients with acute bleeding status
* Hemoglobin concentration below 10g/dL
* Disease directly affecting hematopoiesis (eg. Leukemia, myeloma, aplastic anemia)
* Uncompensated liver cirrhosis, acute hepatitis, alcoholics
* Patients who participated in other clinical studies that could affect prognosis
* Patients who cannot understand the informed consent (eg. Foreigner)

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient older than 20 years and undergong elective valvular heart surgery.
Sampling Method: Probability Sample
Enrollment: 150 (Actual)
Dates: Start 2022-06-23 (Actual); Primary Completion 2024-11-15 (Actual); Study Completion 2025-09-15 (Actual)

PRIMARY OUTCOMES:
Change of hemoglobin concentration level after surgery in patients undergoing heart valve surgery | immediate after surgery, POD1, POD2, POD7, first outpatient vist after discharge (until 6 months)
  Compare the change of hemoglobin concentration level after surgery in patients undergoing heart valve surgery, by dividing the groups according to the level of erythroferron immediately after surgery. The amount of change will be compared based on the lowest level of hemoglobin during the time point after surgery. Since investigators planed to compare the recovery rate as well as the amount of recovery at each time point, investigators planed to record the change of hemoglobin at each time point based on the lowest hemoglobin level after surgery.

SECONDARY OUTCOMES:
Change in serum erythropoietin (EPO) level | From baseline (preoperative) to 6 months postoperatively
  Serum erythropoietin concentration will be measured using a quantitative ELISA assay and reported as mIU/mL. Changes in EPO level from baseline to 6 months will be compared among ERFE tertile groups.
Change in serum hepcidin level | From baseline (preoperative) to 6 months postoperatively
  Serum hepcidin concentration will be measured using liquid chromatography-mass spectrometry (LC-MS) and reported as ng/mL.
Change in hemoglobin (Hb) concentration | From baseline (preoperative) to 6 months postoperatively
  Hemoglobin will be measured using an automated hematology analyzer and reported as g/dL.

CONTACTS AND LOCATIONS:
Locations (1):
- Yonsei University Health System, Severance Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No